CLINICAL TRIAL: NCT01482494
Title: Detection of Pompe Disease in Adult Patients With Myopathies of Uncertain Origin or With Asymptomatic Hyper-CK-emia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jordi Perez Lopez (Other)
Collaborators: Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor-Investigator, Jordi Perez Lopez, Médico Adjunto especialista en Medicina Interna.Responsable de la Unidad de Enfermedades Minoritarias, Hospital Vall d'Hebron
Organization: Hospital Vall d'Hebron (Other)
Other Study IDs: GZ-2011-10784
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Pompe Disease
Keywords: Myopathies; Pompe disease; Polymyositis; Respiratory Insufficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II; Muscular Diseases; Polymyositis; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pompe suspected patients: Patients who go to an Internal Medicine clinic for examination of a limb-girdle myopathy.
  Patients with asymptomatic hyper-CK-emia. Patients with a prior diagnosis of polymyositis. Patients with a myopathy of uncertain origin and respiratory insufficiency. Patients with polymyositis unresponsive to steroid therapy

SUMMARY:
The adult onset form can occur between the second and sixth decades of life as a form of proximal myopathy, predominantly in the pelvic girdle area. Sometimes the first symptoms are shortness of breath and diaphragm weakness which herald progressive proximal muscle weakness. The heart and liver are not affected.

Serum CK (Creatine Kinase) activity is 2 to 10 times higher than normal. EMG (electromyogram) testing usually reveals a myopathic pattern and muscle biopsy may show vacuoles containing an accumulation of glycogen that is not broken down.

Until fairly recently, an assay of acid maltase activity using cultured fibroblasts after biopsy of skin or muscle tissue was required for diagnosis, as leukocytes contain a renal isoenzyme that is not absent in these patients and which can mask the deficit and result in false negatives. In recent years this problem has ben solved by the introduction of acarbose, an inhibitor of renal α-glucosidase; it is also used in the dried blood spot method, which measures acid maltase activity using maltose and acarbose as inhibitors and 4-methylumbelliferyl-D-glucopyranoside as substrate.

DETAILED DESCRIPTION:
Lysosomal storage disorders are inborn errors of metabolism characterized by defects in lysosomal function. Lysosomes contain acid hydrolases whose function is to break down complex molecules in the cell into simpler ones. A deficiency in the activity of any of these enzymes results in the progressive accumulation of substances that cause a storage disease.

Pompe disease is a progressive muscle disease that is often fatal, caused by a deficiency of lysosomal alpha glucosidase (also known as acid maltase) activity. This leads to the accumulation of glycogen in many tissues, most notably in skeletal and cardiac tissues and in muscle tissue. It is therefore also a glycogen storage disease (type II).

It is inherited in an autosomal recessive manner and was the first lysosomal storage disease to be identified. The incidence rate varies by geographic area and ethnic group, and is estimated to be between 1/300,000 to 1:40,000.

It has a broad clinical spectrum that varies with respect to age of onset, rate of progression and extent of organ involvement.

The adult onset form can occur between the second and sixth decades of life as a form of proximal myopathy, predominantly in the pelvic girdle area. Sometimes the first symptoms are shortness of breath and diaphragm weakness which herald progressive proximal muscle weakness. The heart and liver are not affected.

Serum CK (Creatine Kinase) activity is 2 to 10 times higher than normal. EMG (electromyogram) testing usually reveals a myopathic pattern and muscle biopsy may show vacuoles containing an accumulation of glycogen that is not broken down.

Until fairly recently, an assay of acid maltase activity using cultured fibroblasts after biopsy of skin or muscle tissue was required for diagnosis, as leukocytes contain a renal isoenzyme that is not absent in these patients and which can mask the deficit and result in false negatives. In recent years this problem has ben solved by the introduction of acarbose, an inhibitor of renal α-glucosidase; it is also used in the dried blood spot method, which measures acid maltase activity using maltose and acarbose as inhibitors and 4-methylumbelliferyl-D-glucopyranoside as substrate.

Diagnosis is based on clinical suspicion, determination of lysosomal acid alpha-glucosidase activity and confirmation of a mutation in the gene for this enzyme, located on chromosome 17.

Glycogenosis type II is a multisystem disorder and therefore requires a multidisciplinary approach for its treatment. Motor recovery, ventilatory support and nutritional management in patients with gastrointestinal involvement, are seen as fundamental to the treatment. Since 2.000, enzyme replacement therapy with alpha-alglucosidase has been used, whose safety and effectiveness, especially in childhood, has been published in several papers.

ELIGIBILITY:
Inclusion Criteria:

Patients who go to an Internal Medicine clinic for examination of a limb-girdle myopathy.

Patients with asymptomatic hyper-CK-emia. Patients with a prior diagnosis of polymyositis. Patients with a myopathy of uncertain origin and respiratory insufficiency. Patients with polymyositis unresponsive to steroid therapy

Exclusion Criteria:

Patients in treatment Patients with Pompe Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospectively, patients who go to an Internal Medicine clinic for suspected limb-girdle myopathy or patients with asymptomatic hyper-CK-emia shall be included.
  Retrospectively, patients with a prior diagnosis of polymyositis and patients with a myopathy of uncertain origin accompanied by respiratory insufficiency shall be included.
  Before being included in the study, all patients will be asked to give informed consent.
  Acid maltase activity shall be determined by tests performed on leukocytes obtained from peripheral blood samples (5 mL).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico de Barcelona, Barcelona, Barcelona, Spain